CLINICAL TRIAL: NCT06986460
Title: Low Frequency Right Dorsolateral Pre Frontal Cortical Repetitive TMS for Bipolar Depression
Acronym: FLARE
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tyler Kaster (Other)
Collaborators: The Poul Hansen Family Centre for Depression (Unknown); Toronto Western Hospital, Canada (Unknown); University Health Network (UHN) (Unknown)
Responsible Party: Sponsor-Investigator, Tyler Kaster, Principal Investigator, Centre for Addiction and Mental Health
Organization: Centre for Addiction and Mental Health (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4957
Record Dates: First submitted 2025-05-15; First posted 2025-05-23 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Bipolar Depression Depressed Phase
Keywords: rTMS; Bipolar Depression; treatment-resistant; LFR
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Intervention Model Description: Single arm, open label trial to determine if 1Hz rTMS, delivered to the right DLPFC results in a significant reduction of depressive symptoms for individuals with a treatment-resistant bipolar disorder depressive episode (BD-DE) who have not previously responded in the TRIBE study (CTO#: 4343).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low frequency (1Hz) rTMS to the Right Dorsolateral Prefrontal Cortex (Experimental): Individuals will all receive 30 treatments of low frequency (1Hz) rTMS delivered to the Right Dorsolateral Prefrontal Cortex. rTMS treatment will be delivered using the MagPro X100/R30 stimulator and use the Cool-B70 coil (MagVenture, Farum, Denmark), a figure 8 coil with active cooling.
  Interventions: Device: MagPro X100/R30 stimulator, Cool-B70 coil

INTERVENTIONS:
Device: MagPro X100/R30 stimulator, Cool-B70 coil — 1Hz rTMS delivered to the right DLPFC

SUMMARY:
The purpose of this trial is to conduct an adequately powered clinical trial of once daily LFR for individuals diagnosed with treatment-resistant BD-DE who have not responded to iTBS or sham treatment applied to the left DLPFC. This work will develop the evidence supporting the use of LFR rTMS for individuals with treatment-resistant BD-DE who currently have limited treatment options to alleviate their suffering. Participants will come for 30 days of LFR, with a 6-week follow-up period. Symptoms of depression (for determining treatment efficacy) and mania (for determining treatment safety) will be assessed using the 17-item Hamilton Rating Scale for Depression (HRSD-17) and the Young Mania Rating Scale (YMRS) every five treatments during the treatment course, and at 1 week and 6 week after treatment completion.

ELIGIBILITY:
Inclusion Criteria:

1. Must be deemed to have capacity to provide informed consent;
2. Must be an outpatient;
3. Have a DSM 5 diagnosis of bipolar disorder (type I or II), current episode depressed confirmed by Mini-International Neuropsychiatric Interview version 7.0.2 (MINI) assessed during TRIBE trial participation with no contradictory evidence that the current episode is depressed from FLARE trial screening assessments (YMRS>10/PHQ-9 <10);
4. older than 18 years;
5. failure to achieve a clinical response within the TRIBE study (CTO#: 4343) defined as ≤50% response from baseline to 6 weeks on the HRSD-17.
6. Score ≥10 on PHQ-9 at both (i) the 6 weeks follow-up in the TRIBE trial and (ii) at screening;
7. ≤3 months from completion of the TRIBE study;
8. not currently experiencing a mixed or manic episode (YMRS ≤10);
9. no increase or initiation of psychotropic medication with intention of treating depressive symptoms in the 4 weeks prior to screening. This excludes targeted treatment of insomnia with trazodone, melatonin, low-dose doxepin [3-6mg], low-dose benzodiazepines [≤2mg lorazepam daily equivalent], non-benzodiazepine benzodiazepine receptor agonists, or orexin antagonists;
10. currently receiving treatment with one of the following non-anticonvulsant mood stabilizer with evidence for prevention of mania: lithium, quetiapine, asenapine, aripiprazole, paliperidone (>6mg), risperidone, olanzapine, ziprasidone, haloperidol, clozapine (lurasidone and cariprazine are excluded due to lack of evidence for preventing mania);
11. able to adhere to the treatment schedule;
12. pass the TMS adult safety screening questionnaire.

Exclusion Criteria:

1. have a history of MINI diagnosis of a substance use disorder (other than nicotine and/or caffeine) within the last 3 months;
2. have a concomitant major unstable medical illness;
3. have active suicidal intent;
4. are pregnant or intend to get pregnant during the study;
5. have a lifetime MINI diagnosis of schizophrenia or schizoaffective disorder;
6. have psychotic symptoms within the current episode;
7. have a MINI anxiety disorder, trauma-related disorder, obsessive compulsive disorder, or personality disorder assessed by a study investigator to be primary and/or causing greater impairment than BD-DE;
8. failure of an adequate acute course of ECT as defined by ATHF-SF during the current episode;
9. have any clinically significant neurological disorder (e.g., recent major cerebrovascular accident), or any history of seizure except those therapeutically induced by ECT or with clear precipitant (e.g., febrile seizure of childhood, alcohol withdrawal, etc.);
10. have any intracranial implant (e.g., aneurysm clips, shunts, stimulators,) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed;
11. if participating in psychotherapy, must have been in stable treatment for at least 3 months prior to entry into the study, with no anticipation of change in the frequency of therapeutic sessions, or the therapeutic focus over the duration of the study;
12. have a clinically significant laboratory abnormality, in the opinion of the one of the principal investigators;
13. are currently taking lorazepam ≥2 mg daily (or equivalent) due to the potential to limit rTMS efficacy;
14. are currently taking, any dose of an anticonvulsant due to the potential to limit rTMS efficacy;
15. if anticonvulsants have been discontinued prior to screening, at least 5 half-lives have elapsed until screening to allow sufficient drug clearance;
16. have a non-correctable clinically significant sensory impairment (i.e., cannot hear well enough to cooperate with interview).
17. participant was withdrawn from the TRIBE study due to safety concerns or at the discretion of the PI.
18. any history of substance use in the last 4 weeks which poses a safety concern to undergo rTMS as assessed by the PI's review of responses to the trial's 'Substance Use Screening Questions Form'.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-05-27 (Estimated); Primary Completion 2030-05 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Change on the 17-item Hamilton Rating Scale for Depression (HRSD-17) | 6 weeks
  Our primary analysis will be observational, and will calculate the change of the HRSD-17 score from baseline to completion of treatment (i.e., 6 weeks) as the primary outcome. Our primary analysis will be a student's paired t-test to compare the change from baseline to after 6 weeks of treatment with alpha set to 0.05. We will also report the standardized difference to determine the magnitude of change from baseline to completion of treatment.

SECONDARY OUTCOMES:
Symptoms of hypomania/mania | 6 weeks
  Our secondary analysis will also be observational, and will calculate the change of the YMRS score from baseline to completion of treatment (i.e., 6 weeks) as a secondary outcome. Our primary analysis will be a student's paired t-test to compare the change from baseline to after 6 weeks of treatment with alpha set to 0.05. We will also report the standardized difference to determine the magnitude of change from baseline to completion of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Tyler Kaster, Principal Investigator — CAMH
Locations (2):
- Canada (2):
  - University Health Network Toronto Western Hospital, Toronto, Ontario
  - Centre For Addiction and Mental Health (CAMH), Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No
No sharing of IPD, only de-identified. However, we are using ICES databases and not sure how this may apply.